CLINICAL TRIAL: NCT04304131
Title: Colorectal Cancer Screening Using Stool DNA-based SDC2 Methylation Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Collaborators: Genomictree, Inc. (Industry)
Responsible Party: Principal Investigator, Suk-Hwan Lee, Professor, Kyung Hee University Hospital at Gangdong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Earlytect
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Colon Polyp; Healthy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Colorectal cancer (Experimental): Confirmed colorectal cancer under colonoscopy
  Interventions: Diagnostic Test: Earlytect Colon Cancer
- Colon polyp (Experimental): Confirmed colorectal polyp under colonoscopy
  Interventions: Diagnostic Test: Earlytect Colon Cancer
- Healthy (Active Comparator): Confirmed no cancer nor polyp under colonoscopy
  Interventions: Diagnostic Test: Earlytect Colon Cancer

INTERVENTIONS:
Diagnostic Test: Earlytect Colon Cancer — A diagnostic device measuring syndecan 2 methylation status in stool DNA to detect colorectal cancer

SUMMARY:
A study of colorectal cancer screening using stool DNA-based SDC2 methylation test

ELIGIBILITY:
Inclusion Criteria:

* Patient who agreed the clinical trial and signed informed consent
* High risk patient for colorectal cancer (family history of colorectal cancer, history of adenomatous polyp excision, inflammatory bowel disease > 15 years, or history of hereditary colorectal cancer)
* Patient who scheduled to receive colonoscopy
* Stool > 20g before bowel preparation for colonoscopy

Exclusion Criteria:

* No high risk patient under 60 years
* History of colorectal cancer
* Stool < 20g or sample after bowel preparation
* Diarrhea or liquid stool which cannot be evaluated
* Patient who is judged as not suitable for clinical trial including a psychiatric disorder by a physician

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1210 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
SDC2 methylation in stool DNA | 1 year
  positive ratio of SDC2 methylation
sensitivity and specificity of EarlyTect | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Hwan Lee, MD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong; Chang Woo Kim, MD, PhD, Study Director — Ajou University School of Medicine
Locations (8):
- South Korea (8):
  - Busan Hangun Hospital, Busan
  - Koo Hospital, Daegu
  - Severance Hospital, Yonsei University College of Medicine, Seoul
  - Kyung Hee University Hospital at Gangdong, Kyung Hee University School of Medicine, Seoul
  - Dea Hang Hospital, Seoul
  - Eunpyeong St. Mary's Hospital, Seoul
  - Seoul Songdo Hospital, Seoul
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Result] Baylin SB, Ohm JE. Epigenetic gene silencing in cancer - a mechanism for early oncogenic pathway addiction? Nat Rev Cancer. 2006 Feb;6(2):107-16. doi: 10.1038/nrc1799. PMID 16491070
- [Result] Ushijima T. Detection and interpretation of altered methylation patterns in cancer cells. Nat Rev Cancer. 2005 Mar;5(3):223-31. doi: 10.1038/nrc1571. PMID 15719030
- [Result] Laird PW. The power and the promise of DNA methylation markers. Nat Rev Cancer. 2003 Apr;3(4):253-66. doi: 10.1038/nrc1045. PMID 12671664
- [Result] Oh T, Kim N, Moon Y, Kim MS, Hoehn BD, Park CH, Kim TS, Kim NK, Chung HC, An S. Genome-wide identification and validation of a novel methylation biomarker, SDC2, for blood-based detection of colorectal cancer. J Mol Diagn. 2013 Jul;15(4):498-507. doi: 10.1016/j.jmoldx.2013.03.004. Epub 2013 Jun 7. PMID 23747112
- [Result] Xue M, Lai SC, Xu ZP, Wang LJ. Noninvasive DNA methylation biomarkers in colorectal cancer: A systematic review. J Dig Dis. 2015 Dec;16(12):699-712. doi: 10.1111/1751-2980.12299. PMID 26565661
- [Result] Mansour H. Cell-free nucleic acids as noninvasive biomarkers for colorectal cancer detection. Front Genet. 2014 Aug 27;5:182. doi: 10.3389/fgene.2014.00182. eCollection 2014. PMID 25221563
- [Result] Oh TJ, Oh HI, Seo YY, Jeong D, Kim C, Kang HW, Han YD, Chung HC, Kim NK, An S. Feasibility of quantifying SDC2 methylation in stool DNA for early detection of colorectal cancer. Clin Epigenetics. 2017 Dec 4;9:126. doi: 10.1186/s13148-017-0426-3. eCollection 2017. PMID 29225717
- [Result] Han YD, Oh TJ, Chung TH, Jang HW, Kim YN, An S, Kim NK. Early detection of colorectal cancer based on presence of methylated syndecan-2 (SDC2) in stool DNA. Clin Epigenetics. 2019 Mar 15;11(1):51. doi: 10.1186/s13148-019-0642-0. PMID 30876480
- [Derived] Kim CW, Kim H, Kim HR, Won DD, Nam WJ, Min BS, Oh TJ, An S, Lee SH. A Stool DNA-Based SDC2 Methylation Test for the Early Detection of Colorectal Cancer in an Asymptomatic, High-Risk Population: A Multicenter Prospective Randomized Trial. Am J Gastroenterol. 2025 Mar 1;120(3):614-622. doi: 10.14309/ajg.0000000000003044. Epub 2024 Aug 21. PMID 39292188
- [Derived] Kim CW, Kim H, Kim HR, Kye BH, Kim HJ, Min BS, Oh TJ, An S, Lee SH. Colorectal cancer screening using a stool DNA-based SDC2 methylation test: a multicenter, prospective trial. BMC Gastroenterol. 2021 Apr 15;21(1):173. doi: 10.1186/s12876-021-01759-9. PMID 33858326